CLINICAL TRIAL: NCT07322965
Title: Evaluation of the Effect of BRUDYGLAUCO (DHA + Citicoline) in Patients With Glaucoma
Brief Title: Evaluation of BRUDYGLAUCO (DHA + Citicoline) in Patients With Glaucoma
Acronym: BRUDYGLAUCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Catala de Retina (Other)
Collaborators: Hospital de la Esperanza (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICR-02-24
Record Dates: First submitted 2025-03-25; First posted 2026-01-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Glaucoma; Primary Open Angle Glaucoma (POAG); Neuroprotection
Keywords: glaucoma; Primary Open-Angle Glaucoma (POAG); Neuroprotection; Visual Field; DHA (Docosahexaenoic Acid); Citicoline; Nutritional Supplement; Clinical Trial; Randomized Controlled Trial (RCT); Visual Function
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, parallel-group study. Participants will be randomly assigned in a 1:1 ratio to receive either BrudyGlauco (DHA + Citicoline) or a placebo for 12 months. The study will evaluate changes in visual function, treatment safety, and adherence. The study design ensures that neither participants nor investigators know the assigned treatment group, minimizing bias
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study in which both participants and investigators are masked to treatment. The placebo and BrudyGlauco capsules are identical in appearance and packaging to maintain blinding. The treatment assignment is known only to the unmasked study coordinator and the designated data manager responsible for randomization. Blinding will be maintained until the final analysis, except in cases where unblinding is necessary for patient safety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BrudyGlauco (Experimental): Participants receive BrudyGlauco (DHA + Citicoline) orally, taking two capsules at lunchtime for 12 months.
  Interventions: Dietary Supplement: BrudyGlauco
- Placebo Group (Placebo Comparator): Participants receive placebo (sunflower oil capsules) orally, taking two capsules at lunchtime for 12 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: BrudyGlauco — Participants in the experimental group will receive BrudyGlauco, a dietary supplement containing docosahexaenoic acid (DHA) and citicoline.
  Arms: BrudyGlauco
Dietary Supplement: Placebo — Participants in the placebo comparator group will receive identical-looking capsules containing sunflower oil.
  Arms: Placebo Group

SUMMARY:
This study aims to evaluate the effects of BrudyGlauco, a nutritional supplement containing DHA (docosahexaenoic acid) and citicoline, on visual function in people with glaucoma. Glaucoma is a progressive optic neuropathy that can lead to vision loss. Current treatments focus on lowering eye pressure, but there are other pathogenic factors and the use of additional therapies that could protect or regenerate the optic nerve would be beneficial.

This is a randomized, double-blind, placebo-controlled, and multicenter clinical trial. Participants will be randomly assigned to receive either BrudyGlauco or a placebo for 12 months. The study will assess changes in visual field, safety, and treatment adherence.

The trial is being conducted at the Institut Català de Retina (ICR) and Hospital de la Esperanza. Participants will undergo regular eye exams, visual field tests, and follow-ups to monitor potential improvements in visual function.

The results of this study will help determine if BrudyGlauco can provide neuroprotective benefits for people with glaucoma and improve their quality of life.

DETAILED DESCRIPTION:
This study investigates the potential neuroprotective or neuromodulatory effects of BrudyGlauco, a nutritional supplement containing docosahexaenoic acid (DHA) and citicoline, in patients with glaucoma. Glaucoma is a progressive optic neuropathy that leads to visual field deterioration and, in severe cases, to blindness. Although current treatments primarily target intraocular pressure (IOP), the progression of vision loss in glaucoma could benefit by therapies aimed at protecting the optic nerve.

This randomized, double-blind, placebo-controlled trial will assess the effects of BrudyGlauco on visual function over 12 months, with the primary outcome focusing on changes in visual field function. Secondary outcomes include treatment safety, tolerance, and the persistence of any observed effects after treatment discontinuation.

Participants will be recruited from Institut Català de Retina (ICR) and Hospital de la Esperanza, where they will undergo regular ophthalmologic evaluations. These evaluations include visual field tests to measure any changes in vision and DHA biomarker analysis using the Dry Blood Spot (DBS) method to assess DHA levels in erythrocyte membranes.

An interim analysis at six months will allow for an early assessment of efficacy and safety. The final results will determine whether BrudyGlauco has neuroprotective potential for glaucoma management, offering insights into its ability to protect the optic nerve and potentially improve quality of life for patients living with the disease.

Glaucoma is one of the leading causes of blindness worldwide, and current treatments that focus on lowering IOP are not always sufficient to prevent the progressive loss of vision. This study will explore whether DHA and citicoline, known for their neuroprotective properties, can offer additional benefits beyond traditional treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic glaucoma (primary or secondary, open-angle or closed-angle) diagnosed in at least one eye, meeting the following criteria:

   Structural damage: Thinning of the neuroretinal rim, peripapillary hemorrhage, or reduction in the nerve fiber layer, confirmed by OCT or color fundus photography.

   Functional damage: At least 3 contiguous abnormal points outside the 95% confidence limit in the pattern deviation map of the visual field.
2. At least 4 reliable visual field (VF) tests before study enrollment.
3. Age between 50 and 75 years.
4. If both eyes meet the inclusion criteria, the eye with the worst Mean Deviation (MD) will be selected as the study eye.

Exclusion Criteria:

1. Use of any vitamin or nutraceutical supplement in the month prior to screening.
2. Any condition that could alter visual field testing, including:

   Neurological diseases. Retinal diseases. Advanced cataracts. Treatment with Lyrica (Pregabalin) due to its effect on visual fields.
3. Hypersensitivity to acetylsalicylic acid (aspirin) (cross-reactivity risk with citicoline).
4. Ocular surgery or laser treatment in the 3 months prior to enrollment or planned during the study.
5. Mean Deviation (MD) of the visual field worse than -20 dB or better than -3 dB.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in visual function assessed by Mean Deviation (MD) at 12 months | 12 months
  Change from baseline in visual function assessed by Mean Deviation (MD) at 12 months
Change from baseline in visual function assessed by Visual Field Index (VFI) at 12 months | 12 months
  Change from baseline in visual function assessed by Visual Field Index (VFI) at 12 months

SECONDARY OUTCOMES:
Rate of change (slope) in Visual Field Index (VFI) before, during, and after treatment | Baseline, 6 months, 12 months, and 3 months post-treatment (15 months total)
  Rate of change (slope) in Visual Field Index (VFI) before, during, and after treatment
Rate of change (slope) in Mean Deviation (MD) before, during, and after treatment | Baseline, 6 months, 12 months, and 3 months post-treatment (15 months total).
  Rate of change (slope) in Mean Deviation (MD) before, during, and after treatment
Incidence of treatment-emergent adverse events during BrudyGlauco treatment | 12 months
  Incidence of treatment-emergent adverse events during BrudyGlauco treatment
Change from baseline in Visual Field Index (VFI) at 6 months | 6 months
  Change from baseline in Visual Field Index (VFI) at 6 months
Incidence of adverse events at 6 months | 6 months
  Incidence of adverse events at 6 months
Change in Mean Deviation (MD) 3 months after treatment discontinuation | 3 months post-treatment (15 months total).
  Change in Mean Deviation (MD) 3 months after treatment discontinuation
Change in Visual Field Index (VFI) 3 months after treatment discontinuation | 3 months post-treatment (15 months total).
  Change in Visual Field Index (VFI) 3 months after treatment discontinuation

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Institut Català de Retina, Barcelona, Barcelona
  - Hospital del Mar | Centre Esperança, Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No